CLINICAL TRIAL: NCT01390233
Title: Comparison of Pre-Induction Cervical Ripening Using Prepidil Gel Administered Through a Urinary Balloon Catheter.
Brief Title: Comparison of Pre-Induction Cervical Ripening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-60
Record Dates: First submitted 2011-02-11; First posted 2011-07-08 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Failed Labour
Keywords: Labor, obstetric; Labor, induced
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Urinary Balloon Catheter Only (Active Comparator): A urinary balloon catheter will be placed through the cervix into the lower uterine segment and the bulb inflated with 40ml of saline. The catheter will be taped to the patient's thigh and placed under traction using a liter bag of saline. The catheter will be deflated and removed after 6 hours. If spontaneously expelled from the uterus, time of expulsion will be noted. Six hours after insertion of catheter, a digital exam will be performed and Bishop score recorded. If no active labor at time of catheter removal or expulsion, standardized protocol of oxytocin will commence. Labor management will be at the discretion of the physician.
  Interventions: Device: Urinary Balloon Catheter
- Prepadil Only (Active Comparator): Prepidil Only : Prepidil gel will be inserted into the vaginal fornix according to manufacturer's direction. No oxytocin or other intervention will commence until 6 hours after insertion of gel. Six hours after insertion of gel, digital exam will be performed and Bishop score recorded. If no active labor 6 hours after the administration of gel, standardized protocol of oxytocin will commence. Labor management will be at the discretion of the physician.
  Interventions: Drug: Prepidil Gel
- Combined Urinary Catheter & Prepidil Gel (Experimental): A urinary balloon catheter will be placed through the cervix into the lower uterine segment and the bulb inflated with 40ml of saline. The catheter will be taped to the patient's thigh and placed under traction using a liter bag of saline. Prepidil gel will be inserted through the catheter into the lower uterine segment, in a dose equivalent to manufacturer's recommendation. No oxytocin or other intervention will commence until 6 hours after insertion of the catheter and administration of prepidil gel (even if catheter is spontaneously expelled). After 6 hours, digital exam will be performed and Bishop score recorded. If no active labor, standardized protocol of oxytocin will commence.
  Interventions: Other: Combined Urinary Catheter & Prepidil Gel

INTERVENTIONS:
Drug: Prepidil Gel — Pre-induction cervical ripening using dinoprostone gel in the vagina.
  Arms: Prepadil Only
Device: Urinary Balloon Catheter — Pre-induction cervical ripening using a urinary balloon catheter device.
  Other Names: Foley Catheter
  Arms: Urinary Balloon Catheter Only
Other: Combined Urinary Catheter & Prepidil Gel — Pre-induction cervical ripening using dinoprostone gel injected through a urinary balloon catheter placed in the lower uterine segment.
  Other Names: Foley catheter; Prepidil Gel
  Arms: Combined Urinary Catheter & Prepidil Gel

SUMMARY:
This study is designed to assess the effectiveness of a combination method of induction of labor using a urinary balloon catheter and prostaglandin gel.

The vaginal delivery rate for medical induction of labor is lower than the vaginal delivery rate for spontaneous labor. As a consequence, the frequency of cesarean section for failed induction in the United States is rising. This has led to a renewed effort to examine the effectiveness of the varied methods of induction.

The study is a randomized, unblinded trial of urinary balloon catheter and prostaglandin gel for induction of labor in term pregnant patients. Pregnant women presenting to the Palmetto Health Richland for a scheduled induction of labor will be offered enrollment in the trial. Patients who enroll in the study will be randomized into one of 3 study arms: urinary balloon catheter only, prostaglandin gel only and combination urinary balloon catheter and prostaglandin gel. Randomization will be per sealed envelope from the locked nurse medication storage area (Pyxis) located in Labor and Delivery at Palmetto Health Richland. The investigator will be given the next sequentially numbered study randomization envelope by the patient's nurse. The randomization assignment will be unblinded to the patient and her physicians. If the patient is not in active labor 6 hours after initiation of the intervention, a standardized protocol of oxytocin will commence. Labor management will be at the discretion of the physician.

DETAILED DESCRIPTION:
Title: Comparison of pre-induction cervical ripening using Prepidil gel administered through a urinary balloon catheter

Precis- This study is designed to assess the effectiveness of a combination method of induction of labor using a urinary balloon catheter and prostaglandin gel.

Background

Induction of labor is a common intervention during pregnancy1. The frequency of hospital admissions for induction of labor is increasing in the United States. Indications for induction of labor include maternal disease, fetal complications and social/geographical issues. Obstetricians may also choose elective induction, to facilitate delivery at term for the physician or patient who does not have a medical indication for delivery.

The vaginal delivery rate for medical induction of labor is lower than the vaginal delivery rate for spontaneous labor. As a consequence, the frequency of cesarean section for failed induction in the United States is rising2. This has led to a renewed effort to examine the effectiveness of the varied methods of induction3-5.

The vaginal delivery rate for induction of labor can be predicted by assessing the patient's cervical examination prior to induction. The Bishop Score uses the cervical examination components to predict the vaginal delivery rate for a particular patient. A low or poor Bishop score predicts a low success rate for vaginal delivery.

There are 3 common methods used to induce labor. The first are physiological methods such as breaking the patient's water or causing contractions by nipple stimulation. Breaking the patient's water requires a high (favorable) Bishop Score and cannot be safely performed with a low (poor) Bishop score. This method has a higher success rate in patients who have had a prior vaginal delivery. Nipple stimulation has been associated with an increased risk of tachysystole (too frequent contractions) and non-reassuring fetal heart rate patterns. It is not considered an acceptable method of induction in the United States.

Physical methods include pre-induction cervical ripening with laminaria or urinary balloon catheter6. Both of these methods are designed to force the cervix to open mechanically. Laminaria are small sticks of dehydrated seaweed which are placed in the cervical canal. As the sticks hydrate, the cervical canal dilates. Balloon urinary catheters are inserted into the cervical canal. The balloon is inflated in the lower uterine segment. A weight is placed on the catheter to apply traction which forces the fluid-filled balloon to dilate the cervical canal. Urinary balloon catheters have been used alone7,8, with saline infusion9-11 or with prostaglandin infusion12-16.

Pharmacological methods include ergot alkaloids, prostaglandin E and F series and oxytocin. Ergot alkaloids cause forceful uterine contractions and have been used to treat postpartum hemorrhage. Ergot alkaloids may cause severe hypertension during induction of labor and are not used in the United States. Prostaglandin E and F series cause increased uterine muscle tone (tonic contractions). They are used for pre-induction cervical ripening. The different prostaglandins have varying complications which may include nausea, vomiting, diarrhea and fever. Use of misoprostol for pre-induction cervical ripening has been associated with an increased risk of uterine rupture both in normal patients and in patients who have had previous cesarean sections17. The method of drug delivery for prostaglandin medications has varied. It can be administered as an oral tablet, a vaginal suppository, a vaginal gel, or by infusion into the lower uterine segment via a urinary balloon catheter. It is unclear, based on evidence-based medicine, whether any particular method of delivery is superior to another. The Food and Drug Administration of the United States (FDA) has approved the use of Prepidil gel (prostaglandin E2) for pre-induction cervical ripening18,19. Prepidil gel is administered as a gel into the vaginal fornix using a syringe. Oxytocin is a pituitary hormone which can be used to augment spontaneous labor or to induce labor. It results in both increased uterine tone (tonic contractions) and increased contraction frequency (clonic contractions). It is considered the most physiologic method of pre-induction cervical ripening. Oxytocin is administered by intravenous infusion.

Methods of induction can be used individually or in combination. The most common combination method for induction of labor is the use of prostaglandin for pre-induction cervical ripening followed by oxytocin.

Objectives-

The current study is a randomized, unblinded trial of urinary balloon catheter and prostaglandin gel for induction of labor in term pregnant patients. The primary outcome to be studied is vaginal delivery rate for urinary balloon catheter alone, prostaglandin gel alone and a combination of urinary balloon catheter and prostaglandin gel. Secondary outcomes to be studied include the safety of the method, composite maternal morbidity and composite neonatal morbidity.

The null hypothesis is that there is no difference in the vaginal delivery rate between the three study protocols.

Study Design and Methods-

Pregnant women presenting to the Palmetto Health Richland for a scheduled induction of labor will be offered enrollment in the trial.

Eligible patients will undergo an interview with the investigator. Enrollment pre-requisites and exclusions will be reviewed with the patient. The patient will also be provided with written information regarding the safety of prepidil as an pre-induction cervical ripening agent and the safety of urinary balloon catheters as a pre-induction cervical ripening agent. The investigator will review general information on the trial and an informed consent. Patients who decline enrollment in the trial will have the method of pre-induction cervical ripening chosen by their physician.

Inclusion Criteria:

1. Single, live fetus
2. Cephalic (head-first) presentation
3. Reassuring fetal health assessment
4. Gestational age between 26 and 42 weeks
5. Maternal age 18 and above
6. Bishop score less than 5

Exclusion Criteria:

1. Multiple Gestation (twins, triplets, quadruplets)
2. Fetal demise
3. Fetal malpresentation
4. Estimated fetal weight less than 500 grams or more than 4000 grams
5. Placenta previa
6. Non-reassuring fetal health assessment
7. Maternal asthma
8. Latex allergy
9. Spontaneous labor
10. Other contraindication to vaginal delivery

Patients who enroll in the study will be randomized into 3 study arms: urinary balloon catheter only, prostaglandin gel only and combination urinary balloon catheter and prostaglandin gel. Randomization will be made by choosing a sealed envelope from the locked nurse medication storage area (Pyxis) located on Labor and Delivery at Palmetto Health Richland. Randomization will be 1:1:1 with randomization envelopes prepared by statisticians at the University of South Carolina Arnold School of Public Health. The investigator will be given the next sequentially numbered study envelope by the patient's nurse. The randomization included will be unblinded to the patient and her physicians.

URINARY BALLLOON CATHETER ONLY ARM

The patient will be placed in the lithotomy position, either in the bed or in stirrups. A baseline digital exam of the cervix will be performed by the physician and a Bishop score recorded. A urinary balloon catheter will be placed through the cervix into the lower uterine segment, either digitally or with the aid of a speculum. Once the catheter is properly positioned, the bulb will be inflated with 40ml of normal saline. The urinary balloon catheter will then be secured to the patient's thigh using tape. The catheter will then be placed under traction by attaching it to a liter bag of saline.

The catheter will be deflated and removed after 6 hours, with the time of removal recorded in the medical record. If the catheter is spontaneously expelled from the uterus, the time of expulsion will be noted by the nurse. Six (6) hours after insertion of the catheter, the physician will perform a digital cervical exam and a Bishop score recorded.

If the patient is not in active labor at the time of catheter removal or expulsion, a standardized protocol of oxytocin will commence. Labor management will be at the discretion of the physician. Artificial rupture of membranes may also be carried out at the physician's discretion.

PREPIDIL ONLY ARM

The patient will be placed in the lithotomy position, either in the bed or in stirrups. A baseline digital exam of the cervix will be performed by the physician and a Bishop score recorded in the medical record.

Prepidil gel will be inserted into the vaginal fornix according to the manufacturer's direction. No oxytocin or other intervention will commence until 6 hours after insertion of the gel. Six (6) hours after insertion of the gel, the physician will perform a digital cervical exam and a Bishop score recorded.

If the patient is not in active labor 6 hours after the administration of Prepidil gel, a standardized protocol of oxytocin will commence. Labor management will be at the discretion of the physician. Artificial rupture of membranes may also be carried out at the physician's discretion.

COMBINED URINARY BALLOON CATHETER AND PREPIDIL GEL ARM

The patient will be placed in the lithotomy position, either in the bed or in stirrups. A baseline digital exam of the cervix will be performed by the physician and a Bishop score recorded. A urinary balloon catheter will be placed through the cervix into the lower uterine segment, either digitally or with the aid of a speculum. Once the catheter is properly positioned, the bulb will be inflated with 40ml of normal saline. The urinary balloon catheter will then be secured to the patient's thigh using tape. The catheter will then be placed under traction by attaching it to a liter bag of saline.

Prepidil gel will be inserted through the urinary balloon catheter into the lower uterine segment, in a dose equivalent to the manufacturer's recommendation. No oxytocin or other intervention will commence until 6 hours after insertion of the catheter and prepidil gel (even if the catheter is spontaneously expelled prior to that time). Six (6) hours after insertion of the catheter and gel, the physician will perform a digital cervical exam and a Bishop score recorded.

The catheter will be deflated and removed after 6 hours, with the time of removal noted by the nurse. If the catheter is spontaneously expelled from the uterus, the time of expulsion will be noted by the nurse. If the patient is not in active labor 6 hours after insertion of prepidil gel, a standardized protocol of oxytocin will commence. Labor management will be at the discretion of the physician. Artificial rupture of membranes may also be carried out at the physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Single, live fetus
2. Cephalic (head-first) presentation
3. Reassuring fetal health assessment
4. Gestational age between 26 and 42 weeks
5. Maternal age 18 and above
6. Bishop score less than 5

Exclusion Criteria:

1. Multiple Gestation (twins, triplets, quadruplets)
2. Fetal demise
3. Fetal malpresentation
4. Estimated fetal weight less than 500 grams or more than 4000 grams
5. Placenta previa
6. Non-reassuring fetal health assessment
7. Maternal asthma
8. Latex allergy
9. Spontaneous labor
10. Other contraindication to vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-07; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul C Browne, MD, Principal Investigator — University of South Carolina
Locations (1):
- Palmetto Health Richland Hospital, Columbia, South Carolina, United States

REFERENCES:
- [Background] Menacker F, Hamilton BE. Recent trends in cesarean delivery in the United States. NCHS Data Brief. 2010 Mar;(35):1-8. PMID 20334736
- [Background] Greybush M, Singleton C, Atlas RO, Balducci J, Rust OA. Preinduction cervical ripening techniques compared. J Reprod Med. 2001 Jan;46(1):11-7. PMID 11209625
- [Background] Matonhodze BB, Hofmeyr GJ, Levin J. Labour induction at term--a randomised trial comparing Foley catheter plus titrated oral misoprostol solution, titrated oral misoprostol solution alone, and dinoprostone. S Afr Med J. 2003 May;93(5):375-9. PMID 12830603
- [Background] Kelly AJ, Malik S, Smith L, Kavanagh J, Thomas J. Vaginal prostaglandin (PGE2 and PGF2a) for induction of labour at term. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD003101. doi: 10.1002/14651858.CD003101.pub2. PMID 19821301
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] Heinemann J, Gillen G, Sanchez-Ramos L, Kaunitz AM. Do mechanical methods of cervical ripening increase infectious morbidity? A systematic review. Am J Obstet Gynecol. 2008 Aug;199(2):177-87; discussion 187-8. doi: 10.1016/j.ajog.2008.05.005. PMID 18674661
- [Background] James C, Peedicayil A, Seshadri L. Use of the Foley catheter as a cervical ripening agent prior to induction of labor. Int J Gynaecol Obstet. 1994 Dec;47(3):229-32. doi: 10.1016/0020-7292(94)90566-5. PMID 7705527
- [Background] Cromi A, Ghezzi F, Tomera S, Uccella S, Lischetti B, Bolis PF. Cervical ripening with the Foley catheter. Int J Gynaecol Obstet. 2007 May;97(2):105-9. doi: 10.1016/j.ijgo.2006.10.014. Epub 2007 Feb 20. PMID 17316649
- [Background] Saunders JR. Foley-catheter induction of labour. Br Med J. 1972 Oct 28;4(5834):237. doi: 10.1136/bmj.4.5834.237-a. No abstract available. PMID 5082574
- [Background] Hemlin J, Moller B. Extraamniotic saline infusion is promising in preparing the cervix for induction of labor. Acta Obstet Gynecol Scand. 1998 Jan;77(1):45-9. PMID 9492717
- [Background] Karjane NW, Brock EL, Walsh SW. Induction of labor using a foley balloon, with and without extra-amniotic saline infusion. Obstet Gynecol. 2006 Feb;107(2 Pt 1):234-9. doi: 10.1097/01.AOG.0000198629.44186.c8. PMID 16449106
- [Background] Wagman H, Usherwood M. Intrauterine death treated with intrauterine extra-amniotic prostaglandin E2. Br J Clin Pract. 1974 Sep;28(9):318. PMID 4464977
- [Background] Luengo J, Keirse MJ, Bennebroek Gravenhorst J. Extraamniotic prostaglandin F2 alpha for intrauterine death and fetal abnormality. Eur J Obstet Gynecol Reprod Biol. 1977;7(5):325-9. doi: 10.1016/0028-2243(77)90017-x. PMID 299460
- [Background] Fuchs AR, Goeschen K, Rasmussen AB, Rehnstrom JV. Cervical ripening and plasma prostaglandin levels. Comparison of endocervical and extra-amniotic PGE2. Prostaglandins. 1984 Aug;28(2):217-27. doi: 10.1016/0090-6980(84)90058-3. PMID 6594722
- [Background] Liu HS, Chang YK, Chu TY, Yu MH, Chen WH. Extra-amniotic balloon with PGE2 versus extra-ovular Foley catheter with PGF2alpha in mid-trimester pregnancy termination. Int J Gynaecol Obstet. 1998 Oct;63(1):51-4. doi: 10.1016/s0020-7292(98)00114-3. PMID 9849711
- [Background] Sherman DJ, Frenkel E, Pansky M, Caspi E, Bukovsky I, Langer R. Balloon cervical ripening with extra-amniotic infusion of saline or prostaglandin E2: a double-blind, randomized controlled study. Obstet Gynecol. 2001 Mar;97(3):375-80. doi: 10.1016/s0029-7844(00)01168-6. PMID 11239640
- [Background] American College of Obstetricians and Gynecologists Committee on Obstetric Practice. ACOG Committee Opinion No. 342: induction of labor for vaginal birth after cesarean delivery. Obstet Gynecol. 2006 Aug;108(2):465-8. doi: 10.1097/00006250-200608000-00045. PMID 16880321
- [Background] ACOG Committee Opinion. American College of Obstetrician and Gynecologist. ACOG Committee Opinion. Number 283, May 2003. New U.S. Food and Drug Administration labeling on Cytotec (misoprostol) use and pregnancy. Obstet Gynecol. 2003 May;101(5 Pt 1):1049-50. doi: 10.1016/s0029-7844(03)00396-x. PMID 12738178
- [Background] Thomas IL, Chenoweth JN, Tronc GN, Johnson IR. Preparation for induction of labour of the unfavourable cervix with Foley catheter compared with vaginal prostaglandin. Aust N Z J Obstet Gynaecol. 1986 Feb;26(1):30-5. doi: 10.1111/j.1479-828x.1986.tb01524.x. PMID 3524549
- [Background] St Onge RD, Connors GT. Preinduction cervical ripening: a comparison of intracervical prostaglandin E2 gel versus the Foley catheter. Am J Obstet Gynecol. 1995 Feb;172(2 Pt 1):687-90. doi: 10.1016/0002-9378(95)90594-4. PMID 7856707
- [Background] Orhue AA. Induction of labour at term in primigravidae with low Bishop's score: a comparison of three methods. Eur J Obstet Gynecol Reprod Biol. 1995 Feb;58(2):119-25. doi: 10.1016/0028-2243(94)01963-0. PMID 7774736
- [Background] Ghezzi F, Massimo F, Raio L, Di Naro E, Balestreri D, Bolis P. Extra-amniotic Foley catheter and prostaglandin E(2) gel for cervical ripening at term gestation. Eur J Obstet Gynecol Reprod Biol. 2001 Aug;97(2):183-7. doi: 10.1016/s0301-2115(00)00544-3. PMID 11451546
- [Background] Sciscione AC, Nguyen L, Manley J, Pollock M, Maas B, Colmorgen G. A randomized comparison of transcervical Foley catheter to intravaginal misoprostol for preinduction cervical ripening. Obstet Gynecol. 2001 Apr;97(4):603-7. doi: 10.1016/s0029-7844(00)01186-8. PMID 11275035
- [Background] Chung JH, Huang WH, Rumney PJ, Garite TJ, Nageotte MP. A prospective randomized controlled trial that compared misoprostol, Foley catheter, and combination misoprostol-Foley catheter for labor induction. Am J Obstet Gynecol. 2003 Oct;189(4):1031-5. doi: 10.1067/s0002-9378(03)00842-1. PMID 14586350
- [Background] Niromanesh S, Mosavi-Jarrahi A, Samkhaniani F. Intracervical Foley catheter balloon vs. prostaglandin in preinduction cervical ripening. Int J Gynaecol Obstet. 2003 Apr;81(1):23-7. doi: 10.1016/s0020-7292(02)00392-2. PMID 12676389
- [Background] Al-Taani MI. Comparison of prostaglandin E2 tablets or Foley catheter for labour induction in grand multiparas. East Mediterr Health J. 2004 Jul-Sep;10(4-5):547-53. PMID 16335645
- [Background] Afolabi BB, Oyeneyin OL, Ogedengbe OK. Intravaginal misoprostol versus Foley catheter for cervical ripening and induction of labor. Int J Gynaecol Obstet. 2005 Jun;89(3):263-7. doi: 10.1016/j.ijgo.2005.02.010. Epub 2005 Apr 2. PMID 15919393
- [Background] Dalui R, Suri V, Ray P, Gupta I. Comparison of extraamniotic Foley catheter and intracervical prostaglandin E gel for preinduction cervical ripening. Acta Obstet Gynecol Scand. 2005 Apr;84(4):362-7. doi: 10.1111/j.0001-6349.2005.00662.x. PMID 15762966
- [Background] Owolabi AT, Kuti O, Ogunlola IO. Randomised trial of intravaginal misoprostol and intracervical Foley catheter for cervical ripening and induction of labour. J Obstet Gynaecol. 2005 Aug;25(6):565-8. doi: 10.1080/01443610500231450. PMID 16234141
- [Background] Adeniji AO, Olayemi O, Odukogbe AA. Intravaginal misoprostol versus transcervical Foley catheter in pre-induction cervical ripening. Int J Gynaecol Obstet. 2006 Feb;92(2):130-2. doi: 10.1016/j.ijgo.2005.10.010. Epub 2005 Dec 2. No abstract available. PMID 16325816
- [Background] Saleem S. Efficacy of dinoprostone, intracervical foleys and misoprostol in labor induction. J Coll Physicians Surg Pak. 2006 Apr;16(4):276-9. PMID 16624192
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264

RESULTS

PARTICIPANT FLOW:
Groups:
- Prepadil Only: Prepidil gel will be inserted into the vaginal fornix according to manufacturer's direction. No oxytocin or other intervention will commence until 6 hours after insertion of gel. Six hours after insertion of gel, digital exam will be performed and Bishop score recorded. If no active labor 6 hours after the administration of gel, standardized protocol of oxytocin will commence. Labor management will be at the discretion of the physician.
  Dinoprostone Gel: Pre-induction cervical ripening using dinoprostone gel in the vagina.
- Combined Urinary Catheter & Prepadil Gel: A urinary balloon catheter will be placed through the cervix into the lower uterine segment and the bulb inflated with 40ml of saline. The catheter will be taped to the patient's thigh and placed under traction using a liter bag of saline. Prepidil gel will be inserted through the catheter into the lower uterine segment, in a dose equivalent to manufacturer's recommendation. No oxytocin or other intervention will commence until 6 hours after insertion of the catheter and administration of prepidil gel (even if catheter is spontaneously expelled). After 6 hours, digital exam will be performed and Bishop score recorded. If no active labor, standardized protocol of oxytocin will commence.
  Urinary Balloon Catheter Device and Dinoprostone Gel: Pre-induction cervical ripening using dinoprostone gel injected through a urinary balloon catheter placed in the lower uterine segment.
Period: Overall Study
Arm/Group | Urinary Balloon Catheter Only | Prepadil Only | Combined Urinary Catheter & Prepadil Gel
Started | 35 | 31 | 36
Completed | 30 | 29 | 30
Not Completed | 5 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Urinary Balloon Catheter Only | Prepadil Only | Combined Urinary Catheter & Prepadil Gel | Total
Number analyzed (Participants) | 34 | 31 | 36 | 101
Age, Continuous [Mean (Full Range); unit: years] | 25 [18 to 37] | 25 [18 to 38] | 26 [18 to 44] | 25 [18 to 44]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 31 | 36 | 101
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 31 | 36 | 101
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 31 | 36 | 101

OUTCOME MEASURES:

1. Primary Outcome: Vaginal Delivery
Description: The primary outcome of this study is vaginal delivery of a liveborn singleton pregnancy. The outcome is considered a vaginal delivery if accomplished by spontaneous vaginal delivery, operative forceps or vacuum forceps. The alternate outcome is delivery by cesarean section.
Time Frame: Gestational age 26-42 weeks
Measure: Number; unit: participants
Arm/Group | Urinary Balloon Catheter Only | Prepadil Only | Combined Urinary Catheter & Prepadil Gel
Number analyzed (Participants) | 34 | 31 | 36
participants | 20 | 21 | 20

ADVERSE EVENTS:
Time Frame: Entire enrollment period (July 2010 to February 2013)
Arm/Group | Urinary Balloon Catheter Only | Prepadil Only | Combined Urinary Catheter & Prepadil Gel
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/31 | 1/36
Other Adverse Events (participants affected / at risk) | 0/35 | 0/31 | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urinary Balloon Catheter Only (N=35) | Prepadil Only (N=31) | Combined Urinary Catheter & Prepadil Gel (N=36)
Placental Abruption (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) — Patient with pregnancy complicated by prematurity and HELLP syndrome underwent induction of labor in this trial. She subsequently had a placental abruption after enrollment and required an emergency cesarean section.

LIMITATIONS AND CAVEATS:
Limits included: patients enrolled who did not meet inclusion criteria (Bishop score too favorable, but recruited by clinician), patients who were enrolled but catheter could not be placed, patient enrolled who ultimately decided to undergo cesarean.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes